CLINICAL TRIAL: NCT06881654
Title: Home Bleaching With 16% Carbamide Peroxide Using Conventional (Soft) Tray or Rigid Tray: a Randomized Blinded Equivalence Clinical Trial.
Brief Title: 16% Carbamide Peroxide Home Bleaching: Soft vs. Rigid Tray in a Randomized Blinded Equivalence Trial
Acronym: Rigid tray
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Isabel Giráldez de Luis, Lecturer PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URJC_IDIBO_3; Research Ethics Committee (Other: Universidad Rey Juan Carlos)
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Tooth Discolouration
Keywords: sensitivity; gingival irritation; comfort; home-bleaching; soft-tray; rigid tray
MeSH Terms: conditions — Tooth Discoloration; Hypersensitivity | interventions — Tooth Bleaching

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOFT-TRAY. Patients in this group will have the whitening gel applied using the splint (Active Comparator): Participants will apply the 16% carbamide peroxide bleaching gel to a 1 mm soft ethylene vinyl acetate tray for 2 hours per day.
- RIGID-TRAY. Patients in this group wear a 0.5 mm rigid tray. (Other): Patients in this group should have the 16% carbamide peroxide bleaching gel applied in a 0.5 mm rigid polyethylene terephthalate tray for 2 hours per day.
  Interventions: Procedure: Bleaching teeth

INTERVENTIONS:
Procedure: Bleaching teeth — Traditionally, home bleaching has been done with soft silicone trays. Patients now wear aligners, which are rigid trays used for orthodontic treatment. The use of rigid trays for home whitening has not been validated. The aim of this clinical trial is to analyse the effectiveness, comfort and sensitivity perceived by patients when whitening with 0.5 mm rigid aligners.
  Arms: RIGID-TRAY. Patients in this group wear a 0.5 mm rigid tray.

SUMMARY:
The aim of this clinical study is to evaluate patient satisfaction, bleaching efficacy, and the risk and severity of tooth sensitivity and gingival irritation during home bleaching with 16% carbamide peroxide using conventional (soft) trays or rigid trays. A total of 100 patients will be selected to undergo home bleaching with either soft or rigid trays (n=50). Bleaching will be performed with 16% carbamide peroxide (Whiteness Perfect 16%, FGM, Joinville, SC, Brazil) for 2 hours daily for 3 weeks (21 days). Patient satisfaction will be assessed initially, weekly during the 3 weeks of treatment, and one month after completion of treatment using a questionnaire based on a visual analogue scale (VAS) from 0 to 10. Tooth colour will be assessed at baseline, 1 and 3 weeks during treatment, and 1, 6 and 12 months after treatment using the VITA Easyshade V spectrophotometer and the VITA Classical and VITA Linearguide 3D-MASTER scales (VITA Zahnfabrik, Bad Säckingen, Germany). The risk and intensity of tooth sensitivity and gingival irritation were recorded in a diary using a 0-10 VAS during treatment. Patient satisfaction data were analysed using Student's paired t-test. Colour change will be compared between groups using Student's t-test. The absolute risk of tooth sensitivity and gingival irritation was compared between groups using Fisher's exact test. Relative risk and confidence intervals (CI) were also calculated. The intensity of dental sensitivity and gingival irritation was analysed using Student's t-test for independent samples. The significance level will be set at 5% for all statistical tests.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to evaluate patient satisfaction, whitening efficacy, and the risk and severity of tooth sensitivity and gingival irritation after home bleaching with 16% carbamide peroxide using conventional (soft) trays or rigid trays. In addition, to assess whether there is a difference in patient satisfaction using a 0-10 visual analogue scale with conventional (soft) splints or rigid splints during home bleaching with 16% carbamide peroxide. To evaluate whether there is a difference in whitening efficacy using the VITA Easyshade V spectrophotometer and the VITA Classical and VITA Linearguide 3D-MASTER scales with conventional (soft) splints or rigid splints during home bleaching with 16% carbamide peroxide. To assess whether there is a difference in the absolute risk and intensity of tooth sensitivity using a visual analogue scale from 0 to 10 when using conventional (soft) splints or rigid splints during home bleaching with 16% carbamide peroxide and finally to assess whether there is a difference in the absolute risk and intensity of gingival irritation using a visual analogue scale from 0 to 10 when using conventional (soft) splints or rigid splints during home bleaching with 16% carbamide peroxide.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with vital teeth without restorations, single crowns, implants and/or bridges on the anterior teeth.
* Absence of dental caries in the teeth to be whitened.
* Patients with satisfactory oral hygiene and periodontal health, not undergoing periodontal maintenance and not using chlorhexidine mouthwashes. Patients with recession and no sensitivity were included.
* The absence of sensitivity was measured by applying air with the syringe of the dental equipment.
* Patients whose canines were at least A2-A3 in colour.

Exclusion Criteria:

* Patients who have already undergone bleaching (less than 5 years).
* Patients undergoing orthodontic treatment.
* Patients with white stains or changes in enamel development or staining.
* Patients with a history of trauma to the anterior teeth.
* Patients requiring internal bleaching.
* Smokers.
* Pregnant or lactating mothers.
* Patients with allergy to any of the bleaching components.
* Patients with oral mucosal changes (desquamative gingivitis, oral lichen planus, leukoplakia, etc.).
* Patients with medical conditions considered by the investigators to compromise the safety of the study or the individual patient.
* Patients with poor oral hygiene.
* Patients with a history of hypersensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-12-17 (Estimated)

PRIMARY OUTCOMES:
Dental Sensitivity Visual Analog Scale (VAS) 0-10 | 1 month
  To assess whether there is a difference in the absolute risk and intensity of tooth sensitivity, using a visual analogue scale of 0 to 10, when using conventional (soft) trays or rigid trays during home bleaching with 16% carbamide peroxide.
Patient's oral quality of life Visual Analog Scale (VAS) 0-10 | 1 month
  To assess whether there is a difference in patient satisfaction using a 0-10 visual analogue scale when using conventional (soft) trays or rigid trays for home bleaching with 16% carbamide peroxide.
Whitening Efficacy CIEL*a*b* | 1 month
  To evaluate whether there is a difference in whitening efficacy using the VITA Easyshade V spectrophotometer and the VITA Classical and VITA Linearguide 3D-MASTER scales when using conventional (soft) trays or rigid trays during home bleaching with 16% carbamide peroxide.
Gingival irritation VAS (0-10) | 1 month
  To assess whether there is a difference in the absolute risk and intensity of gingival irritation using a visual analogue scale of 0 to 10 when using conventional (soft) trays or rigid trays during home bleaching with 16% carbamide peroxide.

CONTACTS AND LOCATIONS:
Overall Officials: LAURA CEBALLOS, PhD Proffesor, Study Chair — Universidad Rey Juan Carlos; Victoria Fuentes, PhD Reader, Study Director — Universidad Rey Juan Carlos; ISABEL GIRALDEZ, PhD Assistan Proffesor, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The patients have signed a consent form in which they give their data to the Universidad Rey Juan Carlos, but not to the entire research community. The results obtained will be shared, but not the personal data of the participants, in accordance with the regulations on the protection of personal data, specifically the European Regulation 679/2016, of 27 April, on General Data Protection, as well as the Organic Law 3/2018, of 5 December, on the Protection of Personal Data and Guarantee of Digital Rights.

REFERENCES:
- [Background] Levrini L, Paracchini L, Bakaj R, Diaconu A, Cortese S. Dental bleaching during orthodontic treatment with aligners. Int J Esthet Dent. 2020;15(1):44-54. PMID 31994535
- [Background] Chagas AS, Freitas KMS, Cancado RH, Valarelli FP, Canuto LFG, Oliveira RCG, Oliveira RCG. Level of satisfaction in the use of the wraparound Hawley and thermoplastic maxillary retainers. Angle Orthod. 2020 Jan;90(1):63-68. doi: 10.2319/031319-197.1. Epub 2019 Jul 22. PMID 31335161
- [Background] Carneiro TS, Favoreto MW, Centenaro GG, Carneiro OS, Crovador CJ, Stanislawczuk R, Reis A, Loguercio AD. Does simultaneous versus individual-arch at-home dental bleaching regimen influence patient satisfaction? A randomized clinical trial. J Esthet Restor Dent. 2022 Dec;34(8):1263-1271. doi: 10.1111/jerd.12962. Epub 2022 Sep 20. PMID 36125103